CLINICAL TRIAL: NCT01966120
Title: A Randomized, Double-blind, Phase III, Multi-center Study to Evaluate the Safety and Efficacy of BF-200 ALA (Ameluz®) Versus Placebo in the Field-directed Treatment of Mild to Moderate Actinic Keratosis With Photodynamic Therapy (PDT) When Using the BF-RhodoLED® Lamp
Brief Title: Safety and Efficacy Study for the Field-directed Treatment of Actinic Keratosis (AK) With Photodynamic Therapy (PDT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biofrontera Bioscience GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALA-AK-CT007; 2013-002510-12 (EudraCT Number)
Record Dates: First submitted 2013-10-17; First posted 2013-10-21 (Estimated); Results first posted 2016-12-19 (Estimated); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Actinic Keratosis
Keywords: Photodynamic Therapy; Field-directed Treatment
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid; Photochemotherapy; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BF-200 ALA gel (Active Comparator): Photodynamic therapy with BF-RhodoLED in combination with BF-200 ALA.
  Interventions: Drug: BF-200 ALA gel; Procedure: Photodynamic therapy with BF-RhodoLED
- Placebo to BF-200 ALA gel (Placebo Comparator): Photodynamic therapy with BF-RhodoLED in combination with a nanoemulsion gel formulation similar to BF-200 ALA, but without the active ingredient 5-aminolevulinic acid.
  Interventions: Drug: Placebo to BF-200 ALA gel; Procedure: Photodynamic therapy with BF-RhodoLED

INTERVENTIONS:
Drug: BF-200 ALA gel — BF-200 ALA was applied over 1-2 fields of approximately 20 cm² in total, allowed to dry for approximately 10 minutes, and covered with occlusive tape material for 3 h.
  Other Names: Ameluz
  Arms: BF-200 ALA gel
Drug: Placebo to BF-200 ALA gel — The reference product was a placebo (a nanoemulsion gel formulation similar to the Investigational Medicinal Product (IMP), but without the active ingredient). The placebo was packaged, assigned to each patient, and administered in the same way as the IMP.
  Arms: Placebo to BF-200 ALA gel
Procedure: Photodynamic therapy with BF-RhodoLED — After cleaning the lesions, the entire treatment field(s) were illuminated using the novel narrow spectrum BF-RhodoLED lamp, a red light illumination source (approximately 635 nm) developed by Biofrontera, until a total light dose of 37 J/cm² (per treated field) was achieved.
  Other Names: PDT

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of BF-200 ALA (Ameluz) versus placebo in the field-directed treatment of mild to moderate actinic keratosis with photodynamic therapy (PDT) when using the BF-RhodoLED lamp.

DETAILED DESCRIPTION:
The study was performed as a randomized, multicentre, double-blind, placebo- controlled, parallel-group, phase III trial with BF-200 ALA and placebo in seven centres in Germany. A total of 94 patients were screened in this study; 87 were randomized (55 patients received BF-200 ALA, 32 received placebo). Patients received one PDT. If residual lesions remained at 3 months after treatment, PDT was repeated. Illumination was performed with the PDT lamp BF-RhodoLED.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 85 years of age (inclusive)
* Presence of 4 to 8 clinically confirmed actinic keratosis (AK) target lesions of mild to moderate intensity within 1-2 fields

Exclusion Criteria:

* History of hypersensitivity to 5-ALA or any ingredient of BF-200 ALA
* Current treatment with immunosuppressive therapy
* Presence of other malignant or benign tumors of the skin within the treatment area (eg malignant melanoma, basal cell carcinoma (BCC) or squamous cell carcinoma (SCC)) within the last 4 weeks
* Confirmed diagnosis of SCC for the representative lesion by screening biopsy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Reinhold, Prof. Dr., Principal Investigator — Dermatologisches Zentrum Bonn
Locations (1):
- Dermatologisches Zentrum Bonn Friedensplatz, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reinhold U, Philipp-Dormston WG, Dirschka T, Ostendorf R, Aschoff R, Berking C, Jager A, Schmitz B, Foguet M, Szeimies RM. Long-term follow-up of a randomized, double-blind, phase III, multi-centre study to evaluate the safety and efficacy of field-directed photodynamic therapy (PDT) of mild to moderate actinic keratosis using BF-200 ALA versus placebo and the BF-RhodoLED(R) lamp. J Eur Acad Dermatol Venereol. 2025 Aug;39(8):1449-1459. doi: 10.1111/jdv.20452. Epub 2024 Dec 12. PMID 39666443

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial was conducted in Germany with 7 study sites (Bonn, Dresden, Munich, Wuppertal, Mönchengladbach, Cologne, and Recklinghausen) who recruited patients.
Pre-assignment Details: 94 patients were screened, 87 patients were randomized (55 patients to BF-200 ALA and 32 patients to placebo) and treated. 7 patients were screening failures: 3 withdrew consent, 2 did not meet the in- /exclusion criteria, and 2 failed for other reasons (recruitment stop).
Groups:
- BF-200 ALA: Photodynamic therapy with BF-200 ALA
  After lesion preparation, the entire content of 1 tube of verum was applied to the treatment fields identified for this study at screening. The verum was applied to the entire field(s) covering a size of approx. 20 cm² with a film of about 1 mm thickness. Application near the eyes, nostrils, mouth, ears, or mucosa was to be avoided (by a distance of 1 cm). After application, the investigational medicinal product (IMP) was allowed to dry for approx. 10 minutes before occlusion.
  Following incubation of 3 hours (+/- 10 minutes) the dressing was removed and the remnant gel wiped off with a 0.9% saline solution. Thereafter illumination was performed using BF-RhodoLED lamp (635 nm) applying a total light dose of 37 J/cm² (per treated field). This treatment was performed once and repeated after 12 weeks if no complete response was observed.
- Placebo to BF-200 ALA: Photodynamic therapy with a nanoemulsion gel formulation similar to BF-200 ALA, but without the active ingredient 5-aminolevulinic acid.
  After lesion preparation, the entire content of 1 tube of verum was applied to the treatment fields identified for this study at screening. The verum was applied to the entire field(s) covering a size of approx. 20 cm² with a film of about 1 mm thickness. Application near the eyes, nostrils, mouth, ears, or mucosa was to be avoided (by a distance of 1 cm). After application, the IMP was allowed to dry for approx. 10 minutes before occlusion.
  Following incubation of 3 hours (+/- 10 minutes) the dressing was removed and the remnant gel wiped off with a 0.9% saline solution. Thereafter illumination was performed using BF-RhodoLED lamp (635 nm) applying a total light dose of 37 J/cm² (per treated field). This treatment was performed once and repeated after 12 weeks if no complete response was observed.
Period: Overall Study
Arm/Group | BF-200 ALA | Placebo to BF-200 ALA
Started | 55 | 32
Completed | 54 | 26
Not Completed | 1 | 6
Not completed — Withdrawal by Subject | 0 | 5
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- BF-200 ALA: Photodynamic therapy with BF-200 ALA
  After lesion preparation, the entire content of 1 tube of verum was applied to the treatment fields identified for this study at screening. The verum was applied to the entire field(s) covering a size of approx. 20 cm² with a film of about 1 mm thickness. Application near the eyes, nostrils, mouth, ears, or mucosa was to be avoided (by a distance of 1 cm). After application, the IMP was allowed to dry for approx. 10 minutes before occlusion.
  Following incubation of 3 hours (+/- 10 minutes) the dressing was removed and the remnant gel wiped off with a 0.9% saline solution. Thereafter illumination was performed using BF-RhodoLED lamp (635 nm) applying a total light dose of 37 J/cm² (per treated field). This treatment was performed once and repeated after 12 weeks if no complete response was observed.
- Total: Total of all reporting groups
Arm/Group | BF-200 ALA | Placebo to BF-200 ALA | Total
Number analyzed (Participants) | 55 | 32 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 4 | 13
  >=65 years | 46 | 28 | 74
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 50 | 29 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 55 | 32 | 87
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 55 | 32 | 87
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 55 | 32 | 87

OUTCOME MEASURES:

1. Primary Outcome: Overall Patient Complete Response 12 Weeks After the Last Photodynamic Therapy (PDT)
Description: All efficacy variables were evaluated for the FAS. The primary efficacy variable was also analyzed for the PP population. All subgroup analyses were carried out for the FAS. Data for size and grade of AK lesions were analyzed using the last observation carried forward (LOCF) approach, affecting the response rates evaluation.
  Due to the small amount of missing data in the study, which did not have any relevant impact on primary results, sensitivity analyses for missing data were not performed.
  The primary efficacy variable was the overall patient complete response 12 weeks after the last PDT. An overall complete responder was defined as a patient in whom all treated actinic keratosis (AK) lesions were cleared (Olsen score of 0) after the last PDT, i.e. after PDT 1 or after PDT 2 if re-treatment was performed.
Time Frame: 12 weeks after PDT 1 or 12 weeks after PDT 2 which might have been necessary because not all lesions were cleared after the first PDT
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BF-200 ALA | Placebo to BF-200 ALA
Number analyzed (Participants) | 55 | 32
percentage of participants | 90.9 [80 to 97] | 21.9 [9.3 to 40]

2. Primary Outcome: Overall Patient Complete Response 12 Weeks After the Last PDT (PP)
Description: All efficacy variables were evaluated for the FAS. The primary efficacy variable was also analyzed for the PP population. All subgroup analyses were carried out for the FAS. Data for size and grade of AK lesions were analyzed using the last observation carried forward (LOCF) approach, affecting the response rates evaluation.
  Due to the small amount of missing data in the study, which did not have any relevant impact on primary results, sensitivity analyses for missing data were not performed.
  The primary efficacy variable was the overall patient complete response 12 weeks after the last PDT. An overall complete responder was defined as a patient in whom all treated AK lesions were cleared (Olsen score of 0) after the last PDT, i.e. after PDT 1 or after PDT 2 if re-treatment was performed.
Time Frame: as for outcome 1
Population: Per Protocol Set (PP)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BF-200 ALA | Placebo to BF-200 ALA
Number analyzed (Participants) | 50 | 27
percentage of participants | 90.0 [78.2 to 96.7] | 25.9 [11.1 to 46.3]

3. Secondary Outcome: Patient Histopathological Confirmed Response Rate
Description: For the secondary confirmatory analysis, several superiority hypotheses were tested within a pre-defined hierarchic multiple testing procedure as described in the Statistical Analysis Protocoll (SAP).
  The key secondary efficacy variables were tested strictly in a pre-defined order to ensure the family-wise error rate (FWER) and the testing procedure had to be stopped once the first non-significant test was obtained.
  The results of the confirmatory analysis are presented in the order pre-defined by the confirmatory testing procedure.
  Assessments of the patient histopathological confirmed response (HCR) rates were based on the results from the biopsy taken 12 weeks after the last PDT from a representative AK lesion selected at screening. If the biopsy result for a patient revealed a residual AK, the patient was considered "not cleared" for the analysis irrespectively of the investigator's clinical assessment.
Time Frame: as for outcome 1
Population: Full Analysis Set (FAS) 6 patients (1 BF-200 ALA and 5 Placebo patients) had a missing evaluation of the second biopsy 12 weeks after PDT.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BF-200 ALA | Placebo to BF-200 ALA
Number analyzed (Participants) | 54 | 27
percentage of participants | 77.8 [64.4 to 88] | 22.2 [8.6 to 42.3]

4. Secondary Outcome: Patient Complete Response 12 Weeks After PDT 1
Description: The second key secondary efficacy variable in the hierarchic test procedure was the patient complete response (complete clearance of all treated AK lesions) assessed at 12 weeks after PDT 1.
Time Frame: 12 weeks after PDT 1
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BF-200 ALA | Placebo to BF-200 ALA
Number analyzed (Participants) | 55 | 32
percentage of participants | 61.8 [47.7 to 74.6] | 9.4 [2 to 25]

5. Secondary Outcome: Lesion Complete Response 12 Weeks After Last PDT
Description: The third key secondary efficacy variable in the hierarchic test procedure was the lesion complete response (completely cleared individual AK lesions) assessed at 12 weeks after last PDT.
Time Frame: as for outcome 1
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: Number of Lesions Analyzed
Arm/Group | BF-200 ALA | Placebo to BF-200 ALA
Number analyzed (Participants) | 55 | 32
Number analyzed (Number of Lesions Analyzed) | 298 | 173
percentage of lesions | 94.3 [91 to 96.6] | 32.9 [26 to 40.5]

6. Secondary Outcome: Patient Partial Response 12 Weeks After Last PDT
Description: The fourth key secondary efficacy variable in the hierarchic test procedure was the patient partial response (defined as complete clearance of at least 75% of treated AK lesions) assessed at 12 weeks after last PDT.
Time Frame: as for outcome 1
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BF-200 ALA | Placebo to BF-200 ALA
Number analyzed (Participants) | 55 | 32
percentage of participants | 94.5 [84.9 to 98.9] | 25 [11.5 to 43.4]

7. Secondary Outcome: Change of Total Lesion Area 12 Weeks After Last PDT
Description: The fifth key secondary efficacy variable in the hierarchic test procedure was the change from baseline in the total lesion area per patient assessed at 12 weeks after last PDT.
Time Frame: as for outcome 1
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: percentage of lesion area change
Arm/Group | BF-200 ALA | Placebo to BF-200 ALA
Number analyzed (Participants) | 55 | 32
percentage of lesion area change | -98.2 (9.65) | -45.5 (42.96)

8. Secondary Outcome: Overall Cosmetic Outcome 12 Weeks After Last PDT for Patients With Sum Score at Baseline of 0 to 3
Description: Study personnel assessed and recorded the skin quality of the treated field(s) at baseline and at the end-of-study visit including skin surface, hyperpigmentation, hypopigmentation, mottled or irregular pigmentation, degree of scarring and atrophy.
  Upon visual examination of the treated field(s), the investigator coded the intensity of each skin parameter on a scale of 0 to 3, where 0 = none, 1 = mild, 2 = moderate, and 3 = severe.
  The cosmetic outcome evaluations were based on the sum score of the skin quality assessment (sum of all ratings for each skin parameter) at the end-of-study visit (Visit 4 or Visit 6, if retreated).
  The outcome was calculated using a 5-point scale ranging from "very good" (0) to "impaired" (4) based on the change of the skin quality assessments compared to baseline (0 = 2 points improvement; 1 = 1 point improvement; 2 = no change; 3 = 1 point worsened; 4 = at least 2 points worsened).
Time Frame: as for outcome 1
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BF-200 ALA | Placebo to BF-200 ALA
Number analyzed (Participants) | 54 | 29
percentage of participants
  Very good | 35.2 [22.7 to 49.4] | 17.2 [5.8 to 35.8]
  Good | 24.1 [13.5 to 37.6] | 13.8 [3.9 to 31.7]
  Satisfactory | 24.1 [13.5 to 37.6] | 20.7 [8 to 39.7]
  Unsatisfactory | 11.1 [4.2 to 22.6] | 27.6 [12.7 to 47.2]
  Impaired | 5.6 [1.2 to 15.4] | 20.7 [8 to 39.7]

9. Secondary Outcome: Overall Cosmetic Outcome 12 Weeks After Last PDT for Patients With Sum Score at Baseline of 1 to 3
Description: as for outcome 8
Time Frame: as for outcome 1
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BF-200 ALA | Placebo to BF-200 ALA
Number analyzed (Participants) | 48 | 26
percentage of participants
  Very good | 39.6 [25.8 to 54.7] | 19.2 [6.6 to 39.4]
  Good | 27.1 [15.3 to 41.8] | 15.4 [4.4 to 34.9]
  Satisfactory | 22.9 [12 to 37.3] | 23.1 [9 to 43.6]
  Unsatisfactory | 6.3 [1.3 to 17.2] | 26.9 [11.6 to 47.8]
  Impaired | 4.2 [0.5 to 14.3] | 15.4 [4.4 to 34.9]

10. Other Pre Specified Outcome: Patient Recurrence Rate in Follow-up (Cumulative)
Description: Cumulative numbers of patients with complete response who showed recurrences 12 months after last treatment (PDT-1 or PDT-2, if re-treated). A patient with complete response was regarded as recurrent if at least one baseline AK lesion recurred during the follow-up (FU). Complete response was achieved if all treated lesions of the patient were cleared 12 weeks after the last treatment (PDT-1 or PDT-2, if re-treated). Lesions that showed recurrence at 6-months (FU1) were also defined as recurrent at 12-months follow-up (FU2).
Time Frame: 12 months after last treatment (PDT-1 or PDT-2, if re-treated)
Population: Full analysis set in follow-up phase (FAS-FUP). Recurrence rate was only analyzed in patients with complete clearance/response 12 weeks after the last treatment (PDT-1 or PDT-2, if re-treated). Complete response was achieved if all treated lesions of the patient were cleared 12 weeks after the last treatment (PDT-1 or PDT-2, if re-treated).
Measure: Count of Participants; unit: Participants
Arm/Group | BF-200 ALA | Placebo to BF-200 ALA
Number analyzed (Participants) | 49 | 7
Participants
  Patients cleared 12 weeks after last PDT with any recurrent baseline AK lesion at 12-months FU | 18 | 1
  Patients cleared 12 weeks after last PDT still completely cleared at 12 months FU | 31 | 6

11. Other Pre Specified Outcome: Lesion Recurrence Rate in Follow-up (Cumulative)
Description: Cumulative recurrence rate in follow-up of baseline AK lesions that were cleared 12 weeks after the last treatment (PDT-1 or PDT-2, if re-treated) and recurred during 12 months follow-up. Lesions that showed recurrence at 6-months (FU1) were also defined as recurrent at 12-months follow-up (FU2).
Time Frame: 12 months after last treatment (PDT-1 or PDT-2, if retreated)
Population: Full analysis set in follow-up phase (FAS-FUP). Lesion recurrence rate was only analyzed in lesions which were cleared 12 weeks after the last treatment (PDT-1 or PDT-2, if re-treated).
Measure: Number; unit: AK lesions
Units Other Than Participants: AK Lesions
Arm/Group | BF-200 ALA | Placebo to BF-200 ALA
Number analyzed (Participants) | 54 | 30
Number analyzed (AK Lesions) | 276 | 52
AK lesions
  Baseline AK lesions cleared 12 weeks after last PDT with recurrence during 12 months FU | 25 | 1
  Baseline AK lesions cleared 12 weeks after last PDT and are still completely cleared at 12 months FU | 251 | 51

12. Other Pre Specified Outcome: Skin Quality in Follow-up (6 Months)
Description: Frequency of skin quality changes in follow-up compared to baseline. Study personnel assessed and recorded the skin quality of the treated field(s) at baseline and at the follow up visit (6 months) including skin surface, hyperpigmentation, hypopigmentation, mottled or irregular pigmentation, degree of scarring and atrophy.
  Upon visual examination of the treated field(s), the investigator coded the intensity of each skin parameter on a scale of 0 to 3, where 0 = none, 1 = mild, 2 = moderate, and 3 = severe.
Time Frame: 6 months after last treatment (PDT-1 or PDT-2, if re-treated)
Population: Full analysis set in follow-up (FAS-FUP), considering only patients with data at 6-months follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | BF-200 ALA | Placebo to BF-200 ALA
Number analyzed (Participants) | 54 | 27
Participants
  Skin surface (roughness/dryness/scaliness): None | 34 | 15
  Skin surface (roughness/dryness/scaliness): Mild | 15 | 9
  Skin surface (roughness/dryness/scaliness): Moderate | 4 | 3
  Skin surface (roughness/dryness/scaliness): Severe | 1 | 0
  Hyperpigmentation (independent of texture change or hypopigmentation): None | 35 | 13
  Hyperpigmentation (independent of texture change or hypopigmentation): Mild | 16 | 10
  Hyperpigmentation (independent of texture change or hypopigmentation): Moderate | 3 | 4
  Hyperpigmentation (independent of texture change or hypopigmentation): Severe | 0 | 0
  Hypopigmentation (independent of texture change or hyperpigmentation): None | 42 | 15
  Hypopigmentation (independent of texture change or hyperpigmentation): Mild | 10 | 9
  Hypopigmentation (independent of texture change or hyperpigmentation): Moderate | 2 | 3
  Hypopigmentation (independent of texture change or hyperpigmentation): Severe | 0 | 0
  Mottled or irregular pigmentation (both hyper- and hypopigmentation: None | 37 | 14
  Mottled or irregular pigmentation (both hyper- and hypopigmentation: Mild | 13 | 9
  Mottled or irregular pigmentation (both hyper- and hypopigmentation: Moderate | 4 | 4
  Mottled or irregular pigmentation (both hyper- and hypopigmentation: Severe | 0 | 0
  Degree of scarring (independent of pigmentary changes): None | 44 | 20
  Degree of scarring (independent of pigmentary changes): Mild | 8 | 5
  Degree of scarring (independent of pigmentary changes): Moderate | 2 | 2
  Degree of scarring (independent of pigmentary changes): Severe | 0 | 0
  Atrophy: None | 48 | 21
  Atrophy: Mild | 4 | 4
  Atrophy: Moderate | 2 | 2
  Atrophy: Severe | 0 | 0

13. Other Pre Specified Outcome: Skin Quality in Follow-up (12 Months)
Description: Frequency of skin quality changes in follow-up compared to baseline. Study personnel assessed and recorded the skin quality of the treated field(s) at baseline and at the follow up visit (12 months) including skin surface, hyperpigmentation, hypopigmentation, mottled or irregular pigmentation, degree of scarring and atrophy.
  Upon visual examination of the treated field(s), the investigator coded the intensity of each skin parameter on a scale of 0 to 3, where 0 = none, 1 = mild, 2 = moderate, and 3 = severe.
Time Frame: 12 months after last treatment (PDT-1 or PDT-2, if re-treated)
Population: Full analysis set in follow-up (FAS-FUP), considering only patients with data at 12-months follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | BF-200 ALA | Placebo to BF-200 ALA
Number analyzed (Participants) | 54 | 26
Participants
  Skin surface (roughness/dryness/scaliness): None | 39 | 15
  Skin surface (roughness/dryness/scaliness): Mild | 14 | 9
  Skin surface (roughness/dryness/scaliness): Moderate | 1 | 2
  Skin surface (roughness/dryness/scaliness): Severe | 0 | 0
  Hyperpigmentation (independent of texture change or hypopigmentation): None | 41 | 16
  Hyperpigmentation (independent of texture change or hypopigmentation): Mild | 13 | 9
  Hyperpigmentation (independent of texture change or hypopigmentation): Moderate | 0 | 1
  Hyperpigmentation (independent of texture change or hypopigmentation): Severe | 0 | 0
  Hypopigmentation (independent of texture change or hyperpigmentation): None | 48 | 18
  Hypopigmentation (independent of texture change or hyperpigmentation): Mild | 6 | 7
  Hypopigmentation (independent of texture change or hyperpigmentation): Moderate | 0 | 1
  Hypopigmentation (independent of texture change or hyperpigmentation): Severe | 0 | 0
  Mottled or irregular pigmentation (both hyper- and hypopigmentation: None | 44 | 19
  Mottled or irregular pigmentation (both hyper- and hypopigmentation: Mild | 9 | 4
  Mottled or irregular pigmentation (both hyper- and hypopigmentation: Moderate | 1 | 3
  Mottled or irregular pigmentation (both hyper- and hypopigmentation: Severe | 0 | 0
  Degree of scarring (independent of pigmentary changes): None | 50 | 23
  Degree of scarring (independent of pigmentary changes): Mild | 4 | 3
  Degree of scarring (independent of pigmentary changes): Moderate | 0 | 0
  Degree of scarring (independent of pigmentary changes): Severe | 0 | 0
  Atrophy: None | 52 | 24
  Atrophy: Mild | 2 | 2
  Atrophy: Moderate | 0 | 0
  Atrophy: Severe | 0 | 0

14. Other Pre Specified Outcome: Patients' Satisfaction in Follow-up (6 Months)
Description: Patients' satisfaction of the overall cosmetic outcome was assessed at 6-months follow-up visit using a 5-point scale, where 0=very good, 1=good, 2=satisfactory, 3=unsatisfactory, and 4=impaired. The lowest rating is the best outcome, the highest rating is the worst outcome.
Time Frame: 6 months after last treatment (PDT-1 or PDT-2, if re-treated)
Population: Full analysis set in follow-up (FAS-FUP), considering only patients with data at 6-months follow-up.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | BF-200 ALA | Placebo to BF-200 ALA
Number analyzed (Participants) | 54 | 27
percentage of patients
  Very good or good | 79.6 [66.5 to 89.4] | 59.3 [38.8 to 77.6]
  Very good | 27.8 [16.5 to 41.6] | 33.3 [16.5 to 54.0]
  Good | 51.9 [37.8 to 65.7] | 25.9 [11.1 to 46.3]
  Satisfactory | 16.7 [7.9 to 29.3] | 25.9 [11.1 to 46.3]
  Unsatisfactory | 3.7 [0.5 to 12.7] | 11.1 [2.4 to 29.2]
  Impaired | 0.0 [0.0 to 6.6] | 3.7 [0.1 to 19.0]

15. Other Pre Specified Outcome: Patients' Satisfaction in Follow-up (12 Months)
Description: Patients' satisfaction of the overall cosmetic outcome was assessed at 12-months follow-up visit using a 5-point scale, where 0=very good, 1=good, 2=satisfactory, 3=unsatisfactory, and 4=impaired. The lowest rating is the best outcome, the highest rating is the worst outcome.
Time Frame: 12 months after last treatment (PDT-1 or PDT-2, if re-treated)
Population: Full analysis set in follow-up (FAS-FUP), considering only patients with data at 12-months follow-up.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | BF-200 ALA | Placebo to BF-200 ALA
Number analyzed (Participants) | 54 | 26
percentage of patients
  Very good or good | 77.8 [64.4 to 88.0] | 69.2 [48.2 to 85.7]
  Very good | 35.2 [22.7 to 49.4] | 26.9 [11.6 to 47.8]
  Good | 42.6 [29.2 to 56.8] | 42.3 [23.4 to 63.1]
  Satisfactory | 18.5 [9.3 to 31.4] | 26.9 [11.6 to 47.8]
  Unsatisfactory | 3.7 [0.5 to 12.7] | 3.8 [0.1 to 19.6]
  Impaired | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 13.2]

ADVERSE EVENTS:
Time Frame: up to 11 months
Description: Adverse Events (AEs) expected to occur as local discomfort were reported via patient questionnaires, local skin reactions expected to occur were to be assessed by the assigned study team, any other AEs were to be reported by the patient or according to the assessment of the investigator.
Arm/Group | BF-200 ALA | Placebo to BF-200 ALA
Serious Adverse Events (participants affected / at risk) | 2/55 | 0/32
Other Adverse Events (participants affected / at risk) | 55/55 | 22/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BF-200 ALA (N=55) | Placebo to BF-200 ALA (N=32)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BF-200 ALA (N=55) | Placebo to BF-200 ALA (N=32)
Application site pain (General disorders) | 53 (162) | 16 (30)
Application site erythema (General disorders) | 51 (76) | 11 (14)
Application site pruritus (General disorders) | 21 (25) | 9 (10)
Application site scab (General disorders) | 20 (26) | 1 (1)
Application site exfoliation (General disorders) | 17 (21) | 1 (1)
Application site oedema (General disorders) | 12 (14) | 1 (1)
Application site vesicles (General disorders) | 6 (6) | 0 (0)
Application site discomfort (General disorders) | 5 (7) | 0 (0)
Application site discharge (General disorders) | 3 (5) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor will review results communications prior to public release and has to approve in order to ensure the adequate reporting of study results. The sponsor can't refuse publication for unfair reasons.